CLINICAL TRIAL: NCT04284436
Title: Study in Parkinson Disease of Exercise Phase 3 Clinical Trial: SPARX3
Brief Title: Study in Parkinson Disease of Exercise
Acronym: SPARX3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Pittsburgh (Other); The Parkinson Study Group (Network)
Responsible Party: Principal Investigator, Daniel Corcos, Professor of Physical Therapy and Human Movement Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01NS113851-01 (NIH)
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Exercise (Experimental): Treadmill exercise 4x per week at 80-85% HRmax.
  Interventions: Behavioral: Treadmill walking
- Moderate Intensity Exercise (Active Comparator): Treadmill exercise 4x per week at 60-65% HRmax.
  Interventions: Behavioral: Treadmill walking

INTERVENTIONS:
Behavioral: Treadmill walking — Treadmill walking 4 days per week for 30 minutes in the target heart rate

SUMMARY:
This study is a Phase 3 multi-site, randomized, evaluator-masked, study of endurance treadmill exercise on changes in the Movement Disorder Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part III score at 12 months among persons with early stage Parkinson disease. 370 participants will be randomly assigned to 2 groups: 1)60-65% HRmax or 2)80-85% HRmax 4 times per week. The primary objective is to test whether the progression of the signs of Parkinson's disease is attenuated at 12 months in among persons who have not initiated medication for Parkinson Disease (PD) when they perform high-intensity endurance treadmill exercise.

DETAILED DESCRIPTION:
This study is a Phase 3 multi-site, randomized, evaluator-masked, study of endurance treadmill exercise on changes in the MDS-UPDRS Part III score at 12 months. 370 persons diagnosed with Parkinson's disease who have not yet initiated dopaminergic therapy, age 40-80, will be randomly assigned to 2 groups: 1)60-65% HRmax or 2)80-85% HRmax 4 times per week. Secondary objectives will test hypotheses related to striatal specific binding ratio (SSBR) at 12 months, MDS-UPDRS Part III score, ambulatory mobility (6-minute walk), daily walking activity (steps), cognition, quality of life, cardiorespiratory fitness, blood-derived biomarkers of inflammation and neurotrophic factors at 12 and 18 months. Tertiary objectives will test hypotheses related to 2 characteristics of ambulation at 12 and 18 months. Exploratory objectives will test hypotheses related to the effects of removing the study support that was provided over 18 months on the sustainability and durability of the exercise effects at 24 months. Approximately 29 sites will enroll participants: 27 sites that cover all geographic regions of the USA and 2 sites in Canada. All sites will have a collaboration between movement disorders and exercise specialists.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic Parkinson Disease based on the modified * United Kingdom (UK) PD brain bank criteria and which are consistent with recent criteria proposed for clinically established early established Parkinson's disease that no longer exclude individuals with a family history of Parkinson's disease.
* Hoehn and Yahr stages less than 3
* Disease duration: less than 3 years since disease diagnosis
* Age 40-80 years
* Positive DaTscan™ SPECT by quantitative readout for idiopathic Parkinson disease.

Exclusion Criteria:

* Currently being treated with PD medications such as levodopa or dopamine receptor agonists, monoamine oxidase-B (MAO-B) inhibitors, amantadine, or anticholinergics.
* Expected to require treatment with medication for PD in the first 6 months of the study.
* Use of any PD medication 60 days prior to the baseline visit including but not limited to levodopa, direct dopamine agonists, amantadine, Rasagiline (Azilect), Selegiline (Eldepryl), Artane (trihexyphenidyl).
* Duration of previous use of medications for PD exceeds 60 days.
* Use of neuroleptics/dopamine receptor blockers for more than 30 days in the year prior to baseline visit, or any use within 30 days of baseline visit
* Presence of known cardiovascular, metabolic, or renal disease or individuals with major signs or symptoms suggestive of cardiovascular, metabolic, or renal disease without medical clearance to participate in the exercise program.
* Uncontrolled hypertension (resting blood pressure >150/90 mmHg)
* Individuals with orthostatic hypotension and standing systolic BP below 100 will be excluded. Orthostatic hypotension (OH) is a reduction of systolic blood pressure of at least 20 mm Hg or diastolic blood pressure of at least 10 mm Hg within 3 minutes of standing.
* Hypo- or hyperthyroidism (TSH <0.5 or >5.0 mU/L), abnormal liver function (AST or ALT more than 2 times the upper limit of normal), abnormal renal function (estimated glomerular filtration rate (eGFR) using the MDRD4 equation or the CKD-EPI equation <45mL/min/1.73m2 ).
* Complete Blood Count (CBC) out of range and physician's judgment that abnormal value is clinically significant.
* Recent use of psychotropic medications (e.g., anxiolytics, hypnotics, benzodiazepines, antidepressants) where dosage has not been stable for 28 days prior to screening.
* Serious illness (requiring systemic treatment and/or hospitalization) within the last 4 weeks.
* Any other clinically significant medical condition, psychiatric condition, drug or alcohol abuse, assessment or laboratory abnormality that would, in the judgment of the investigator, interfere with the subject's ability to participate in the study.
* Montreal Cognitive Assessment (MoCA) score of <24.
* Beck Depression Inventory II (BDI) score > 28, indicating severe depression that precludes ability to exercise. Any subject with such a score will be referred to a PCP or physician for further evaluation and management of depression. Individuals with a BDI-II score of 17-28 will be excluded if any of the following conditions are met: (1) individual is suicidal, (2) is in need of depression treatment modification currently or (3) depressive symptoms likely to interfere with adherence to study protocol. Any subject with such a score will be referred to a PCP or physician for further evaluation and management of depression.
* Individuals who have been exercising at greater than moderate intensity for 120 minutes or more per week consistently over the last 6 months will be excluded. Greater than moderate intensity is defined as a range greater than 60-65% HRmax. These individuals are excluded since their exercise activities are greater than the activities they would experience if they were assigned to the 60-65% treatment group. As such, they would be expected to lose fitness.
* Use of the following within 90 days prior to the DAT neuroimaging screening evaluation: modafinil, armodafinil, metoclopramide, alpha-methyldopa, methylphenidate, reserpine, any amphetamine or amphetamine derivative, or use of buproprion within 8 days prior to the DAT neuroimaging screening evaluation. These can compromise DaTscan™ SPECT.
* Known allergy to iodinated products.
* Known hypersensitivity to DaTscan™ SPECT (either to the active substance of 123I-ioflupane or any of the excipients.
* (For women only) Actively breast-feeding an infant, and/or pregnant, or plan to become pregnant in the next 12 months.
* Other disorders, injuries, diseases, or conditions that might interfere with ability to perform endurance exercises (e.g. history of stroke, respiratory problems, traumatic brain injury, orthopedic injury, or neuromuscular disease).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in motor symptoms of Parkinson disease | 12 months
  Change from baseline in the Movement Disorders Society-Unified Parkinson Disease Rating Scale motor score (Part III). The minimum score on the MDS-UPDRS Part III is 0 and the maximum is 132 with higher scores representing worse motor symptoms.

SECONDARY OUTCOMES:
Change in dopaminergic activity | 12 months
  Change from baseline in the striatal specific binding ratio (SSBR) as measured by dopamine transporter imaging
Change in motor symptoms of Parkinson disease | 18 months
  Change from baseline in the Movement Disorders Society-Unified Parkinson Disease Rating Scale motor score (Part III). The minimum score on the MDS-UPDRS Part III is 0 and the maximum is 132 with higher scores representing worse motor symptoms.
Change in walking capacity | 12 months
  Change from baseline in distance in 6-minute walk
Change in walking capacity | 18 months
  Change from baseline in distance in 6-minute walk
Change in activity | 12 months
  Change from baseline in the number of steps
Change in activity | 18 months
  Change from baseline in the number of steps
Change in cognitive function | 12 months
  Change from baseline in the Montreal Cognitive Assessment (MoCA). MoCA scores range between 0 and 30, with higher scores representing a better outcome.
Change in cognitive function | 18 months
  Change from baseline in the Montreal Cognitive Assessment (MoCA). MoCA scores range between 0 and 30, with higher scores representing a better outcome.
Change in fitness | 12 months
  Change from baseline in maximal oxygen consumption measured with peak oxygen volume
Change in fitness | 18 months
  Change from baseline in maximal oxygen consumption measured with peak oxygen volume
Change in quality of life | 12 months
  Change from baseline in quality of life measured with the Parkinson Disease Questionnaire-39. The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month covering 8 dimensions scored on a 5 point ordinal system (0=never, 4=always). Dimension score = sum of scores of each item in the dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better QoL. Overall score can be summarized in the Parkinson's Disease Summary Index (PDSI) or PDQ-39 Summary Index (PDQ-39 SI).PDSI or PDQ-39 SI = sum of dimension total scores divided by 8.
Change in quality of life | 18 months
  Change from baseline in quality of life measured with the Parkinson Disease Questionnaire-39. The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month covering 8 dimensions scored on a 5 point ordinal system (0=never, 4=always). Dimension score = sum of scores of each item in the dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better QoL. Overall score can be summarized in the Parkinson's Disease Summary Index (PDSI) or PDQ-39 Summary Index (PDQ-39 SI).PDSI or PDQ-39 SI = sum of dimension total scores divided by 8.
Initiation of dopaminergic therapy | 12 months
  Time to initiation of dopaminergic therapy
Change in blood derived marker of inflammation | 12 months
  Change from baseline in C-reactive protein
Change in blood derived marker of inflammation | 18 months
  Change from baseline in C-reactive protein
Change in blood derived marker of neuronal development | 12 months
  Change from baseline in brain derived neurotrophic factor (BDNF)
Change in blood derived marker of neuronal development | 18 months
  Change from baseline in brain derived neurotrophic factor (BDNF)

OTHER OUTCOMES:
Change in stride length | 12 months
  Change in stride length assessed using OPAL movement monitors during the 6 minute walk test
Change in stride length | 18 months
  Change in stride length assessed using OPAL movement monitors during the 6 minute walk test
Change in turning velocity | 12 months
  Change in turning velocity assessed using OPAL movement monitors during the 6 minute walk test
Change in turning velocity | 18 months
  Change in turning velocity assessed using OPAL movement monitors during the 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Corcos, PhD, Principal Investigator — Northwestern University
Locations (25):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Iowa State University, Ames, Iowa
  - Louisiana State University, Baton Rouge, Louisiana
  - Boston University (Charles River Campus), Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health, Columbus, Ohio
  - Kent State University, Kent, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Health San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- University of Alberta, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: Yes
All study data (deidentified) and documentation will be shared with the National Institute of Neurological Disease and Stroke.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18 months after the study end.
Access Criteria: Once the data are in the NINDS data repository, NINDS will be responsible for determining with whom the data are shared. No data will be shared directly from the study data coordinating center.

REFERENCES:
- [Background] Schenkman M, Moore CG, Kohrt WM, Hall DA, Delitto A, Comella CL, Josbeno DA, Christiansen CL, Berman BD, Kluger BM, Melanson EL, Jain S, Robichaud JA, Poon C, Corcos DM. Effect of High-Intensity Treadmill Exercise on Motor Symptoms in Patients With De Novo Parkinson Disease: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):219-226. doi: 10.1001/jamaneurol.2017.3517. PMID 29228079
- [Background] Moore CG, Schenkman M, Kohrt WM, Delitto A, Hall DA, Corcos D. Study in Parkinson disease of exercise (SPARX): translating high-intensity exercise from animals to humans. Contemp Clin Trials. 2013 Sep;36(1):90-8. doi: 10.1016/j.cct.2013.06.002. Epub 2013 Jun 14. PMID 23770108
- [Derived] Patterson CG, Joslin E, Gil AB, Spigle W, Nemet T, Chahine L, Christiansen CL, Melanson E, Kohrt WM, Mancini M, Josbeno D, Balfany K, Griffith G, Dunlap MK, Lamotte G, Suttman E, Larson D, Branson C, McKee KE, Goelz L, Poon C, Tilley B, Kang UJ, Tansey MG, Luthra N, Tanner CM, Haus JM, Fantuzzi G, McFarland NR, Gonzalez-Latapi P, Foroud T, Motl R, Schwarzschild MA, Simuni T, Marek K, Naito A, Lungu C, Corcos DM; SPARX3-PSG Investigators. Study in Parkinson's disease of exercise phase 3 (SPARX3): study protocol for a randomized controlled trial. Trials. 2022 Oct 6;23(1):855. doi: 10.1186/s13063-022-06703-0. PMID 36203214

DOCUMENTS (1):
  • Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT04284436/ICF_003.pdf